CLINICAL TRIAL: NCT06928974
Title: Functional Abdominal Wall Reconstruction in Patients With Prune Belly Syndrome
Brief Title: Functional Abdominal Wall Reconstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Górnośląskie Centrum Zdrowia Dziecka (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017/01/01GCZD
Record Dates: First submitted 2025-04-01; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Prune Belly Syndrome
MeSH Terms: conditions — Prune Belly Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Bilateral Pedicled Vastus Lateralis Muscle Flaps Transposition — Bilateral Pedicled Vastus Lateralis Muscle Flaps Transposition to restore the function of underdeveloped or absent rectus abdomini muscles

SUMMARY:
Assessement of outcomes of functional reconstruction of underdeveloped abdominal muscles with the use od pedicled Vastus Lateralis Muscle flaps.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnoes with Prune Belly Syndrome
* severe underdevelopment of rectus abdomini muscles
* patients who underwent microsurgical bipedicled vastus lateralis muscle flaps transposition
* patient undery 18 y.o.

Exclusion Criteria:

* Patient over the age of 18
* Patients who did not agreed for proposed microsurgical reconstruction of the abdominal wall

Exclusion Criteria: Patient over the age of 18

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients diagnosed with Prune Belly syndrome suffering from symptoms related to abdominal wall insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Electromyography | followup reached 96months
  To assess the proper function of transposed muscles the electromyographic tests were used to assess the proper electroactivity of transposed vastus lateralis muscles. The measured values of amplitude (mV) and conduction velocity(ms) were analyzed.
Motor tests - performance of ''sit-up''-like movement | Followup reached 96 months
  Patients were asked to perform situp-like movement with legs fasetned before surgical transposition of muscles and then 12 months postoperatively. It was assessed in 0/1 manner. 0 - patient not able to do the sit-up, 1 - patient able to do the sit-up

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska Curie Memorial National Cancer Center, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopes RI, Baker LA, Denes FT. Modern management of and update on prune belly syndrome. J Pediatr Urol. 2021 Aug;17(4):548-554. doi: 10.1016/j.jpurol.2021.04.010. Epub 2021 Apr 24. PMID 34016542